CLINICAL TRIAL: NCT03360500
Title: The Effect of Cryotherapy Associated With an Exercise Protocol in Pain Control, Physical Function and Quality of Life in Individuals With Knee Osteoarthritis - Randomized Clinical Trial
Brief Title: Cryotherapy Associated With Exercise in Pain Control and Physical Function in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Lucas Ogura Dantas, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRYO-1234
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis,Knee
Keywords: Osteoarthritis, Knee; Cryotherapy; Exercise; Physiotherapy; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EXERCISE PROTOCOL + CRYOTHERAPY (Experimental): Patients with knee osteoarthritis, both sexes, with age between 40 and 75
  Interventions: Other: EXERCISE PROTOCOL + CRYOTHERAPY
- EXERCISE PROTOCOL (Experimental): Patients with knee osteoarthritis, both sexes, with age between 40 and 75
  Interventions: Other: EXERCISE PROTOCOL
- EXERCISE PROTOCOL + PLACEBO (Placebo Comparator): Patients with knee osteoarthritis, both sexes, with age between 40 and 75
  Interventions: Other: EXERCISE PROTOCOL + PLACEBO

INTERVENTIONS:
Other: EXERCISE PROTOCOL + CRYOTHERAPY — Protocol: The therapeutic exercise protocol was designed according to the recommendations and guidelines of evidence-based practices and specific randomized clinical trials of physical exercise intervention for Knee osteoarthritis.
  The suggested parameters for an adequate prescription of physical exercises include the type, application method, intensity, duration, minimum number of sessions and frequency of exercises.
  Cryotherapy: Crushed ice inside two plastic bags. The positioning of the plastic bags will cover the entire knee surface (Anterior, lateral and posterior region). After the positioning of the ice bags, they will be fixed with an elastic bandage (compression). To protect the skin against frost bites, all the knee surface will be covered with a moistened operative field.
  Arms: EXERCISE PROTOCOL + CRYOTHERAPY
Other: EXERCISE PROTOCOL — Protocol: The therapeutic exercise protocol was designed according to the recommendations and guidelines of evidence-based practices and specific randomized clinical trials of physical exercise intervention for Knee osteoarthritis.
  The suggested parameters for an adequate prescription of physical exercises include the type, application method, intensity, duration, minimum number of sessions and frequency of exercises.
  Arms: EXERCISE PROTOCOL
Other: EXERCISE PROTOCOL + PLACEBO — Protocol: The therapeutic exercise protocol was designed according to the recommendations and guidelines of evidence-based practices and specific randomized clinical trials of physical exercise intervention for Knee osteoarthritis.
  The suggested parameters for an adequate prescription of physical exercises include the type, application method, intensity, duration, minimum number of sessions and frequency of exercises.
  Placebo: Sand inside two plastic bags. The positioning of the plastic bags will cover the entire knee surface (Anterior, lateral and posterior region). After the positioning of the sandbags, they will be fixed with an elastic bandage (compression). All the knee surface will be covered with a moistened operative field.
  Arms: EXERCISE PROTOCOL + PLACEBO

SUMMARY:
The purpose of this study is to verify the effect of cryotherapy associated with an exercise protocol in pain control, function and quality of life in individuals with knee osteoarthritis

DETAILED DESCRIPTION:
The purpose of this study is to verify the effect of cryotherapy associated with an exercise protocol in pain control, function and quality of life in individuals with knee osteoarthritis. This is a randomized controlled clinical trial, double-blinded. Will participate in the study 120 patients with knee osteoarthritis, diagnosed with clinical and radiographic criteria of the American College of Rheumatology, of both sexes, aged between 40 and 75 years. The total number of subjects will be divided randomly into three groups of 40 subjects each. During eight weeks, three times per week, each group will receive one type of intervention: Exercise protocol for knee osteoarthritis + cryotherapy, Exercise protocol for knee osteoarthritis + placebo or Exercise protocol for knee osteoarthritis only. A medical certificate will be requested for all participants, showing the capability of practicing physical activities. Every individual will have the following variables evaluated one day pre- and one day post-intervention process: Pain index (VAS), physical function questionnaires (WOMAC) and quality of life (sf-36 questionnaire). Three physical function tests will also be carried out: the 30s sitting and standing chair, Stair test and fast paced test in 40m. Moreover, participants will perform VAS in every physical function test. A follow-up period will be performed.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosed with knee osteoarthritis based on clinical and radiographic criteria of American College of Rheumatology
* Grade 2 or 3 according to the criteria of Kellgren & Lawrence knee osteoarthritis radiographic examination scale.
* Minimum score of 4 cm in Visual Analogue Scale (total 10 cm)
* Medical prescription, showing that the participant is capable of performing physical activities

Main exclusion Criteria:

* Physical therapy within 3 months prior to the research project
* Corticosteroid injection in the knee (in the previous 6 months)
* Medical condition (cardiorespiratory, neurological and / or musculoskeletal)
* Previous ankle, knee or hip surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (Pain scale): Change values from the pre evaluation to the post evaluation | The first measurement in the pre (First day, first week) and in the post (Last day, last week) evaluation - Full protocol - 12 weeks
  A visual analog scale (VAS) will be applied to measure the pain before and 1 day after the intervention. VAS is a well recognized tool to measure the intensity of pain that visually represents the intensity of pain that the individual believes to present. The scale will be positioned in front of the individual and will have a range of 0 to 10 cm, with 0 being the complete absence of pain and 10, the maximum intensity of pain reported by the individual.

SECONDARY OUTCOMES:
WOMAC questionnaire (Self-administered questionnaire): Change values from the pre evaluation to the post evaluation | The second measurement in the pre (First day, first week) and in the post (Last day, last week) evaluation - Full protocol - 12 weeks
  All volunteers will answer to the questionnaire before and 1 day after the intervention. WOMAC is a self-report questionnaire designed to assess the problems experienced by people with OA of the lower limb. The score for the items is expressed through a Likert scale, where the rating is calculated as: none = 0, low = 25 = 50 moderate, severe = 75 and very severe = 100. The maximum score on each section is expressed as a percentage, with higher scores indicating greater pain, stiffness and physical dysfunction. Each point corresponds to a particular dimension (pain, stiffness and physical function). This questionnaire has been translated and validated for the Portuguese language from Brazil.
36-Item Short Form Survey | The third measurement in the pre (First day, first week) and in the post (Last day, last week) evaluation - Full protocol - 12 weeks
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures.
Fast paced test in 40m test: Change values from the pre evaluation to the post evaluation | The fourth measurement in the pre (First day, first week) and in the post (Last day, last week) evaluation - Full protocol - 12 weeks
  Fast paced walking test that is timed by a distance of 4X10 meters, totaling 40 meters. It is used as a direct measure to correlate the ability to walk fast, short distances. Administered at a distance of 10 meters (demarcated by tapes), a cone is placed 2 meters before the start and 2 meters after the end of each marking. The participant is instructed to walk the 10 meters (from the start marking), turn around in the cone and walk another 10 meters, successively until completing the distance of 40 meters. Time is considered only between the tracks (start and end). The final score is calculated based on the speed of the participant performs the procedure and compared with normative values of healthy adults.
Stair test: Change values from the pre evaluation to the post evaluation | The fifth measurement in the pre (First day, first week) and in the post (Last day, last week) evaluation - Full protocol - 12 weeks
  Test where the participant should go up and down a stair in the shortest possible time. The participant will be positioned in front of the stair, and at the therapeut sign must climb the indicated steps (12 steps), and go down, being able to use the handrail as a security instrument. The height of each stair step will be 20 cm, with a handrail, in an illuminated environment, free of traffic and external distractions. A pre-test is performed to identify the need for safety measures. The final score is calculated based on the time the participant performs the procedure and compared with the normative values available for the test
30 seconds chair stand test: Change values from the pre evaluation to the post evaluation | The sixth measurement in the pre (First day, first week) and in the post (Last day, last week) evaluation - Full protocol - 12 weeks
  All volunteers performed the test before and 1 day after the intervention. The 30 seconds chair stand test is administered using an armless chair, with seat height of about 43cm from the ground. The chair has a rubber for not slipping under its support and is placed against a wall to avoid oscillations. The participant sits in the middle of the chair with the back straight, feet apart, aligned with the shoulder width apart and flat on the floor at an angle slightly behind the knee line. Moreover, to help maintain balance, one foot may be slightly placed ahead of the other and arms crossed against the chest. The test consists of the greatest number of times from a sitting position to a standing over a period of 30 seconds. Thus, it is possible to evaluate a wide range of skill levels with scores ranging from 0, for those who cannot complete a single repetition and values greater than 20 reps for the well prepared individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O Dantas, PhD Student, Principal Investigator — Universidade Federal de Sao Carlos; Julya M Perea, Bachelors, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of Sao Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] French HP, Abbott JH, Galvin R. Adjunctive therapies in addition to land-based exercise therapy for osteoarthritis of the hip or knee. Cochrane Database Syst Rev. 2022 Oct 17;10(10):CD011915. doi: 10.1002/14651858.CD011915.pub2. PMID 36250418
- [Derived] Ogura Dantas L, Serafim Jorge AE, Regina Mendes da Silva Serrao P, Aburquerque-Sendin F, de Fatima Salvini T. Cryotherapy associated with tailored land-based exercises for knee osteoarthritis: a protocol for a double-blind sham-controlled randomised trial. BMJ Open. 2020 Jun 1;10(6):e035610. doi: 10.1136/bmjopen-2019-035610. PMID 32482668